CLINICAL TRIAL: NCT01129245
Title: The Effect of a Non-hormonal Cox-2 Inhibitor (Celebrex) on Ovulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Alison Edelman, Assistant Professor SM.OB/GYN Generalist Division, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: OHSU FAMPLAN SFP3-7
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-05

CONDITIONS: Ovulation; Luteal Development
Keywords: Celebrex; prostoglandin inhibitor; ovulation; emergency contraception
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control cycle (No Intervention): Control menstrual cycle
- Pre-LH surge celecoxib administration (Experimental): Pre-LH surge dosing of celecoxib
  Interventions: Drug: Celebrex; Drug: Placebo
- Post-LH surge celecoxib administration (Experimental): Post-LH surge dosing of celecoxib
  Interventions: Drug: Celebrex; Drug: Placebo

INTERVENTIONS:
Drug: Celebrex — 400 mg PO daily intermittently based on hormone and ultrasound findings
  Other Names: Celecoxib
  Arms: Post-LH surge celecoxib administration; Pre-LH surge celecoxib administration
Drug: Placebo — Placebo identical to celecoxib
  Arms: Post-LH surge celecoxib administration; Pre-LH surge celecoxib administration

SUMMARY:
The purpose of this study is to assess the effect that Celebrex (a COX-2 inhibitor and non-steroidal anti-inflammatory drug) has on ovulation.

DETAILED DESCRIPTION:
A prospective randomized double-blind crossover study of healthy reproductive-aged (18-35 years old) women with regular cycles, not currently using or needing hormonal contraception, were recruited. Women will undergo ovarian ultrasound and serum hormone monitoring during four menstrual cycles (control cycle, treatment cycle 1, washout cycle, treatment cycle 2). Subjects received study drug (oral celecoxib 400 mg or placebo) either 1) once daily starting on cycle day 8 and continuing until follicle rupture or the onset of next menses if follicle rupture did not occur (pre-LH surge dosing) or 2) once daily beginning with the LH surge and continued for 6 days (post-LH surge dosing). Women will be randomly assigned to one of the above treatment schemes and received the other in the subsequent treatment cycle.

This study aims to determine if treatment with a highly selective COX2 inhibitor, celecoxib, would be a more effective agent in terms of causing ovulatory dysfunction. This study also aims to determine whether treatment with celecoxib would adversely affect luteal function.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35
* Currently NOT using hormonal contraception
* Cycle length between 26-34 days
* General good health (specifically no hx of: diabetes, cardiac problems, moderate/severe heart burn (GERD), obesity (BMI > 30), hypertension (BP > 130/80)
* Willing and able to agree to randomization and informed consent
* Willing and able to use a menstrual diary to chart bleeding Serum progesterone > 3 ng/ml (from cycle day 18-25)
* Willing and able to return to clinic for bi-weekly for blood tests and ultrasounds throughout cycles 2, 3 & 5

Exclusion Criteria:

* Diabetes
* Cardiac disease
* Moderate to severe heart burn (or GERD) Obesity (BMI > 30) Hypertension (BP > 130/80)
* Allergy to NSAIDS
* Currently pregnant or trying to conceive
* Polycystic Ovarian Syndrome
* Use of hormonal contraception (participants can use barrier methods, spermicide, female or male sterilization, copper intrauterine device, abstinence, or have female partners

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Edelman, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Result] Edelman AB, Jensen JT, Doom C, Hennebold JD. Impact of the prostaglandin synthase-2 inhibitor celecoxib on ovulation and luteal events in women. Contraception. 2013 Mar;87(3):352-7. doi: 10.1016/j.contraception.2012.07.004. Epub 2012 Aug 16. PMID 22902348
- See also: Author Manuscript — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4040982/

RESULTS

PARTICIPANT FLOW:
Groups:
- PreLH Followed by postLH: Control cycle First, preLH surge dosing of celecoxib and postLH surge dosing of placebo. Followed by, preLH surge dosing of placebo and postLH surge dosing of drug.
- PostLH Followed by preLH: Control cycle First, postLH surge dosing of celecoxib and preLH surge dosing of placebo. Followed by, postLH surge dosing of placebo and preLH surge dosing of drug.
Period: Control Cycle (no Celecoxib or Placebo)
Arm/Group | PreLH Followed by postLH | PostLH Followed by preLH
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Treatment Cycle 1
Arm/Group | PreLH Followed by postLH | PostLH Followed by preLH
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout Cycle
Arm/Group | PreLH Followed by postLH | PostLH Followed by preLH
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Treatment Cycle 2
Arm/Group | PreLH Followed by postLH | PostLH Followed by preLH
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: healthy reproductive-aged women with regular cycles, not currently using or needing hormonal contraception
Groups:
- PreLH/postLH: Control cycle First, preLH surge dosing of celecoxib and postLH surge dosing of placebo. Followed by, preLH surge dosing of placebo and postLH surge dosing of drug.
- PostLH/preLH: Control cycle First, postLH surge dosing of celecoxib and preLH surge dosing of placebo. Followed by, postLH surge dosing of placebo and preLH surge dosing of drug.
- Total: Total of all reporting groups
Arm/Group | PreLH/postLH | PostLH/preLH | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (5.9) | 28.5 (4.9) | 27.4 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic, Caucasian | 9 | 8 | 17
  Other | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Cycles With Ovulation Dysfunction When Taken After Ovulation: Extended Luteal Phase
Description: One cycle corresponds to one participant
Time Frame: 4 cycles (approximately 4 months)
Population: Placebo treatment was not analyzed. This cycle was purely included in the study flow to keep investigators blinded to treatment allocation. It was pre-specified that it would not be analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Control Cycle: Monitoring through ovarian ultrasound and serum hormone levels of menstrual cycle prior to receiving any study treatment in order to insure ovulatory activity.
- Pre-LH Celecoxib: Receive celebrex at pre-determined time in menstrual cycle based on hormone levels and ultrasound results
  Celebrex: 400 mg PO daily intermittently based on hormone and ultrasound findings
- Post-LH Surge Celecoxib: Receive celebrex at pre-determined time in menstrual cycle based on hormone levels and ultrasound results.
  Celebrex: 400 mg PO daily intermittently based on hormone and ultrasound findings
Arm/Group | Control Cycle | Pre-LH Celecoxib | Post-LH Surge Celecoxib
Number analyzed (Participants) | 20 | 20 | 20
Participants | 1 | 6 | 5

2. Secondary Outcome: Peak Hormone Levels
Description: Average serum levels of progesterone (ng/mL) and luteinizing hormone (ng/mL) normalized to days of the luteal phase of menstrual cycle.
Time Frame: 4 cycles (approximately 4 months)
Population: One cycle corresponds to one participant. Placebo treatment was not analyzed. This cycle was purely included in the study flow to keep investigators blinded to treatment allocation. It was pre-specified that it would not be analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Control Cycle | Pre-LH Celecoxib | Post-LH Surge Celecoxib
Number analyzed (Participants) | 20 | 20 | 20
ng/mL
  LH (luteinizing hormone) | 39.7 (25) | 46.2 (28.4) | 42.6 (22.2)
  P (progesterone) | 13.3 (3.3) | 13.5 (3.9) | 12.3 (4.7)

3. Secondary Outcome: Peak Estradiol Level
Description: Average serum levels of estradiol (pg/mL) normalized to days of the luteal phase of menstrual cycle.
Time Frame: 4 cycles (approximately 4 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Control Cycle | Pre-LH Celecoxib | Post-LH Surge Celecoxib
Number analyzed (Participants) | 20 | 20 | 20
pg/mL | 274 (99.6) | 289.4 (124.5) | 282.2 (106.7)

ADVERSE EVENTS:
Groups:
- Pre-LH Celecoxib: Received Celebrex at pre-determined time in menstrual cycle based on hormone levels and ultrasound results.
  Celebrex: 400 mg PO daily intermittently based on hormone and ultrasound findings.
Arm/Group | Control Cycle | Pre-LH Celecoxib | Post-LH Surge Celecoxib
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No